CLINICAL TRIAL: NCT06869876
Title: Ortopod CZ Pilot Study (Total Knee Arthoplasty and Postoperative Delirium Czech Republic
Brief Title: Ortopod CZ Pilot Study
Acronym: ORTOPODCZ
Status: Completed | Type: Observational
Sponsor: Tomas Bata Hospital, Czech Republic (Other)
Responsible Party: Principal Investigator, Klára Nekvindová, Deputy Chief for Science, Teaching, and Research, Tomas Bata Hospital, Czech Republic
Other Study IDs: Č.j: 2025-01
Record Dates: First submitted 2025-03-01; First posted 2025-03-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Delirium (POD); Perioperative Neurocognitive Disorders
Keywords: postoperative delirium; CAM- ICU; ALBA; POBAV; Amnesia Light and Brief Assessment,; screening; cognitive assessment; risk factors; seniors
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total knee arthroplasty: Patients above 65 years old undergoing elective total hip arthroplasty.

SUMMARY:
ORTOPOD PILOT STUDY is a non-randomized, non-interventional clinical study that addresses the issue of perioperative neurocognitive disorder (deterioration of cognitive functions in the preoperative and perioperative period) and its impact on the occurrence of postoperative delirium.

Respondents meeting the entry criteria will undergo elective orthopaedic surgery (total hip arthroplasty) under general or regional anaesthesia.

DETAILED DESCRIPTION:
ORTOPOD PILOT STUDY is a non-randomized, non-interventional clinical study that addresses the issue of perioperative neurocognitive disorder (deterioration of cognitive functions in the preoperative and perioperative period) and its impact on the occurrence of postoperative delirium.

Respondents meeting the entry criteria will undergo elective orthopaedic surgery (total hip arthroplasty) under general or regional anaesthesia. Preoperatively, they will be examined using the ALBA and POBAV tests, which serve for rapid and indicative assessment of cognitive functions. Furthermore, the functional capacity of patients will be assessed using the Clinical Frailty Scale, and depression will be evaluated using the Geriatric Depression Scale (questionnaire).

After the procedure, during hospitalization in the ICU/PACU, screening for postoperative delirium will be conducted using the CAM-ICU tool.

The aim of the pilot study is to verify the methodology and obtain baseline data on the incidence of cognitive dysfunction, depression, and frailty preoperatively, as well as the incidence of postoperative delirium in this group of patients before submitting a grant to AZV ČR. The main research question will be whether preoperative cognitive decline (according to the ALBA and POBAV tests) is associated with the occurrence of postoperative delirium. The second research question will be what percentage of patients with preoperative cognitive deficit (according to the ALBA and POBAV tests) undergo elective total hip arthroplasty. Secondary outcomes will include whether there are differences in the ALBA and POBAV test results before and after surgery (cognitive decline after anesthesia and surgery), whether higher Clinical Frailty Scale scores are associated with the occurrence of postoperative delirium, and whether the results on the Geriatric Depression Scale change preoperatively and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65 years (inclusive)

  * Type of procedure: elective hip replacement (TEP) under general or regional anesthesia
* ASA classification I-III
* Absence of sensory impairment (blindness, deafness, deaf-blindness)

Exclusion Criteria:

* Glasgow Coma Scale of 14 or less
* Limited legal capacity
* Known psychiatric illness with the use of psychiatric medications
* Effect of premedication, psychiatric, and analgesic sedative drugs (at the time of cognitive function testing)
* Active oncological disease
* Chronic use of strong opioids
* Re-operation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: "Respondents meeting the entry criteria will undergo elective orthopedic surgery (total hip replacement) under general or regional anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-25 (Actual)

PRIMARY OUTCOMES:
ALBA - cognitive assessment preoperatively | one week before surgery
  Amnesia Light and Brief Assessment (ALBA) is an ultra-brief and universal cognitive test suitable for assessing cognitive impairment, dementia, and other conditions. Test consists of a one-time encoding of a six-word sentence "Indian summer brings the first morning frost.", sequential demonstration of six gestures and their immediate recall in any order (TEGEST) and finally recall of as many correct words as possible of the original sentence.
  The ALBA score norm for the sum of recalled words and gestures is 6-12 points (at least 50% of the maximum), mild impairment is 4-5 points, and severe impairment is 0-3 points. For more educated individuals (with a high school diploma or more, or 15 years of education or more), the ALBA score norm is 8-12 points..
POBAV - cognitive assessment preoperatively | one week before surgery
  POBAV is an abbreviationof Czech title Picture naming and their recall. The test consists of two parts. The persons are to name each of the 20 picture in one word and remember these picture names. When they finish naming the pictures, then they are asked to recall and write as many picture names as they can during one minute.
  Evaluation of Part 1: After completing the entire test, determine the number of naming errors (images not named at all and incorrectly named). Most older individuals should make a naming error in no more than one image.
  Evaluation of Part 2: The number of correctly recalled images will be determined. The number of errors from the total number of written picture names will be substracted to get the number of correctly recalled image names. Most older individuals should recall 6 or more correct image names, while individuals with a high school diploma should recall 7 image names.
Postoperative CAM-ICU | 0. postoperative day, 1. postoperative day, 2. postoperative day.
  CAM-ICU scale:
  FEATURE 1: Alteration/Fluctuation in Mental Status - Present/not present FEATURE 2: Inattention 1: Alteration/Fluctuation in Mental Status -If number of errors >2 = present /not present FEATURE 3: Altered Level of Consciousness (LOC) - present/not present FEATURE 4: Disorganized Thinking - present/not present
  Features 1 and 2 are both present and either Features 3 or 4 are present:
  Delirium present CAM-ICU is positive, delirium is present
ALBA, POBAV and CAM - ICU | one week before surgery,0. postoperative day, 1. postoperative day, 2. postoperative day.
  The research question is: "Is the reduction in cognitive functions according to the ALBA and POBAV tests associated with the occurrence of postoperative delirium in the Czech Republic?

SECONDARY OUTCOMES:
Clinical frailty scale - assessment preoperatively | one week before surgery
  Clinical frailty scale is a way to summarize the overall level of fitness or frailty of an older adult after they had been evaluated by an experienced clinician.
  Frailty score ranging from 1 (very fit) to 9 (terminally ill).
  1. = very fit
  2. = well
  3. = managing well
  4. = vulnerable
  5. = mildly frail
  6. = moderately frail
  7. = severely frail
  8. = very severely frail
  9. = terminally ill
  Research questions:
  Are higher values of the Clinical Frailty Scale before surgery (values 4, 5, or higher) associated with the occurrence of postoperative delirium in Czech Republic? Are higher values of the Clinical Frailty Scale before surgery (values 4, 5, or higher) associated with the worsening of cognitive functions
Age | one week before surgery
  Age of the patients undergoing elective tottal hip arthroplasty, in years.
ALBA - cognitive assessment postoperatively | 3rd day after surgery
  Amnesia Light and Brief Assessment (ALBA) is an ultra-brief and universal cognitive test suitable for assessing cognitive impairment, dementia, and other conditions. Test consists of a one-time encoding of a six-word sentence "Indian summer brings the first morning frost.", sequential demonstration of six gestures and their immediate recall in any order (TEGEST) and finally recall of as many correct words as possible of the original sentence.
  The ALBA score norm for the sum of recalled words and gestures is 6-12 points (at least 50% of the maximum), mild impairment is 4-5 points, and severe impairment is 0-3 points. For more educated individuals (with a high school diploma or more, or 15 years of education or more), the ALBA score norm is 8-12 points..
POBAV - cognitive assessment postoperatively | 3rd day after surgery
  POBAV is an abbreviationof Czech title Picture naming and their recall. The test consists of two parts. The persons are to name each of the 20 picture in one word and remember these picture names. When they finish naming the pictures, then they are asked to recall and write as many picture names as they can during one minute.
  Evaluation of Part 1: After completing the entire test, determine the number of naming errors (images not named at all and incorrectly named). Most older individuals should make a naming error in no more than one image.
  Evaluation of Part 2: The number of correctly recalled images will be determined. The number of errors from the total number of written picture names will be substracted to get the number of correctly recalled image names. Most older individuals should recall 6 or more correct image names, while individuals with a high school diploma should recall 7 image names.

OTHER OUTCOMES:
Gender | one week before surgery
  Gender of the patient undergoing elective total hip arhroplasty. Women or men.
ASA status preoperatively | one week before surgery
  The American Society of Anesthesiologists (ASA) physical status classification system is a grading system to determine the health of a person before a surgical procedure that requires anesthesia ASA I = a normal healthy patient ASA II = a patient with mild systematic disease ASA III = a patient with severe systematic disease
The Geriatric Depression Scale (GDS) | one week before surgery
  The Geriatric Depression Scale (GDS) is a self-report measure of depression in older adults. Users respond in a "Yes/No" format. Scoring: 0 or 1 point (1 point is awarded for the presence of a depressive symptom). 10 questions indicate depression when answered "Yes," and 5 questions (Nos. 1, 5, 7, 11, 13) indicate depression when answered "No." The questionnaire can thus score a maximum of 15 points.0-5 normal mood, 6-10 mild depression, 11+ severe depression
Education | one week before surgery
  Education of the patients in years.
Duration time of the operation | end of the operation
  Cumulatively in minutes. time will be indicated according to the operating protocol
Blood pressure value during surgery | end of the operation
  Blood pressure values at the beginning and end of the procedure, in mmHg (in anesthesia record).
  Hypotension blood pressure 30% lower than baseline pressure, reported cumulatively in minutes.
Spo2 during surgery | end of the operation
  Value at the beginning and end of the procedure (%), desaturation yes/no (Spo2 94 and less%), duration (in minutes).
Blood loss during surgery | end of the operation
  Blood loss cumulative for the procedure in milliliters.
Blood glucose level during surgery | end of the operation
  Sample of blood glucose level taken as part of standard practice, mmol/l.
Circulatory instability during surgery | end of the operation
  Yes or no. Yes when it is necessary to administer norepinephrine or ephedrine.
Norepinephrine during surgery | end of the operation
  Highest dose of noradrenaline during operation, in µg/kg/min. Total duration of norepinephrine administration during surgery in minutes).
Blood loss after the procedure | 3rd day after operation
  Cumulatively in milliliters, during the CAM-ICU screening period (postoperative day 0, postoperative day 1, postoperative day 2). In case of CAM-ICU positivity, the blood loss assessment continues during the CAM-ICU screening period. Blood loss assessment once a day.
  Evaluated will be amount of transfusion units and , Types of blood derivatives given: Deleukocytized erythrocytes, Prothrombin Complex Concentrate (PCC), Pathogen-inactivated plasma, Fresh frozen plasma, fibrinogen, Platelets from buffy coat mixed deleukocytized in replacement solution.
Postoperative nausea and vomiting | 0. postoperative day
  Yes or no. Assessment 0. postoperative day.
Administered hypnotic or/and anxiolytic | 3rd day after operation
  Yes or no. During the CAM-ICU screening period (postoperative day 0, postoperative day 1, postoperative day 2.
Circulatory instability after the procedure | 3rd day after operation
  Yes or no. Y (yes=when it is necessary to administer norepinephrine). During the CAM-ICU screening period (postoperative day 0, postoperative day 1, postoperative day 2.
Norepinephrine after the procedure | 3rd day after operation
  Highest dose of noradrenaline during the day, in µg/kg/min. Total duration of norepinephrine administration after the procedure (in minutes). During the CAM-ICU screening period (postoperative day 0, postoperative day 1, postoperative day 2).
Necessity of re-operation within 3 days | 3rd day after operation
  Yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Tomas Bata Hospital, Zlín, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium — https://journals.lww.com/ejanaesthesiology/fulltext/2017/04000/european_society_of_anaesthesiology_evidence_based.3.aspx
- See also: TEGEST as promising tool for assessing the risk of perioperative neurocognitive disorders — https://bmcgeriatr.biomedcentral.com/articles/10.1186/s12877-024-05302-9

DOCUMENTS (1):
  • Study Protocol (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT06869876/Prot_000.pdf